CLINICAL TRIAL: NCT01045577
Title: A Double-blind, Placebo-controlled, Randomized, Parallel-group Study to Evaluate the Activity of Oral AB1010 in Adults Patients With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB04029
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Psoriasis
Keywords: Severe Psoriasis; Kinase Inhibitor; Masitinib
MeSH Terms: conditions — Psoriasis | interventions — masitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Masitinib (AB1010) (Active Comparator): Masitinib (AB1010)
  Interventions: Drug: Masitinib
- Placebo mactching masitinib (Placebo Comparator): Placebo matching masitinib
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Masitinib — 6 mg/kg/day
  Arms: Masitinib (AB1010)
Drug: Masitinib — 3 mg/kg/day
  Arms: Masitinib (AB1010)
Drug: Placebo — Placebo matching masitinib (3 mg/kg/day and 6 mg/kg/day)
  Arms: Placebo mactching masitinib

SUMMARY:
A double-blind, placebo-controlled, randomized, parallel-group study to evaluate the activity of oral AB1010 in adults patients with moderate to severe chronic plaque psoriasis

DETAILED DESCRIPTION:
To evaluate the activity of oral AB1010, administered at two dose levels during 12 weeks to patients with moderate to severe chronic plaque psoriasis, assessed on :

i)Body Surface Area (BSA), Psoriasis Area and Severity Index (PASI), Overall Lesion Severity (OLS), Physician's Global Assessment (PGA) and Patient's Global Psoriasis Assessment (PGPA) ii)clinical and biological safety parameters iii) pharmacokinetic profile of AB1010

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 18 to 75 years with chronic plaque psoriasis
* Plaque psoriasis covering ≥ 10% BSA
* Disease duration ≥ 6 months
* PASI ≥ 12.0 at screening

Exclusion Criteria:

* Guttate, erythrodermic or pustular psoriasis as sole or predominant form of the disease
* Clinically significant psoriasis flare during screening or at time of enrollment
* Systemic therapy for psoriasis or systemic immunosuppressive therapy for other indications within 28 days prior to enrollment
* Topical treatment for psoriasis within 14 days prior to enrollment
* Use of CYP3A4 moderate and strong inhibitors within 4 weeks prior to randomization
* Active current bacterial, viral (including hepatitis B and C, HIV, EBV, CMV, herpes zoster, herpes simplex), fungal, mycobacterium, protozoan, or other infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-09; Primary Completion 2006-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in BSA after 12 weeks of treatment | 12 weeks

SECONDARY OUTCOMES:
Percentage change from baseline in PASI score, proportion of patients reaching a 90%, 75% or 50% improvement in PASI score after 12 weeks of treatment; time to and duration of first occurrence in PASI 50, 75 and 90 | 12 weeks
Proportion of patients achieving an OLS rating of Minimal or Clear after 12 weeks | 12 weeks
Percentage change from baseline in PGA and PGPA after 12 weeks of treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul ORTONNE, MD, Principal Investigator — CHU NICE